CLINICAL TRIAL: NCT00730379
Title: A Phase I Study of Ridaforolimus (MK8669) and MK0646 in Patients With Advanced Cancer
Brief Title: A Combination Study With Ridaforolimus (MK8669) and Dalotuzumab (MK0646) in Patients With Advanced Cancer (8669-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-004; 2008_538
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — dalotuzumab

ARMS (1):
- 1 (Experimental): ridaforolimus (MK8669) + dalotuzumab (MK0646)
  Interventions: Drug: Comparator: ridaforolimus + dalotuzumab

INTERVENTIONS:
Drug: Comparator: ridaforolimus + dalotuzumab — Starting dose of oral ridaforolimus is 10 mg/day, QD, for five days. Dose rising up to 40 mg/day, QD for five days. Dose range for intravenous dalotuzumab is 7.5 mg/kg/week, 10 mg/kg/week or 7.5 mg/kg/every 14 days. Dalotuzumab will be given as an IV infusion over 1 or 2 hour(s).

SUMMARY:
This study is being done to find the best tolerated dose of ridaforolimus and dalotuzumab in patients who have advanced cancer and to observe any anti-tumor activity in these patients.

DETAILED DESCRIPTION:
Ridaforolimus (MK8669/AP23573) was also known as deforolimus until May 2009

ELIGIBILITY:
Inclusion Criteria:

* You must have confirmed metastatic or advanced cancer that has not responded to standard therapy or where standard therapy does not exist
* In Part C, patients must have a diagnosis of advanced or metastatic colorectal adenocarcinoma or non-small cell lung cancer, and must have received at least 1 but no more than three prior systemic therapy treatment regimens
* You must be over the age of 18 years old
* You must have a ECOG status performance of 0 or 1
* You must have good organ function
* You must be willing to have skin and/or tumor biopsies

Exclusion Criteria:

* You have had cancer treatment within 4 weeks prior to entering the study or you still have bad side effects from previous therapies
* You have an active infection that requires treatment
* You are HIV positive or have a history of Hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To determine the toxicity profile, maximum tolerated dose and recommended phase II dose. | MTD from Day 1 to Day 28 in Cycle 1 for disease progression

SECONDARY OUTCOMES:
To measure pharmacokinetic and pharmacodynamic parameters with oral ridaforolimus as a single agent and in combination with dalotuzumab | At prescribed timepoints as defined in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Di Cosimo S, Sathyanarayanan S, Bendell JC, Cervantes A, Stein MN, Brana I, Roda D, Haines BB, Zhang T, Winter CG, Jha S, Xu Y, Frazier J, Klinghoffer RA, Leighton-Swayze A, Song Y, Ebbinghaus S, Baselga J. Combination of the mTOR inhibitor ridaforolimus and the anti-IGF1R monoclonal antibody dalotuzumab: preclinical characterization and phase I clinical trial. Clin Cancer Res. 2015 Jan 1;21(1):49-59. doi: 10.1158/1078-0432.CCR-14-0940. Epub 2014 Oct 15. PMID 25320355